CLINICAL TRIAL: NCT06352489
Title: Posterior Component Separation in the Management of the Complex Ventral Hernia
Brief Title: Evaluation of Posterior Component Separation Technique in the Management of Complex Ventral Hernia.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Mohamed Yehya, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Posterior component separation
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCS with TAR (Active Comparator): The posterior component separation technique utilizes the retro-rectus space, accessed by incising the posterior rectus sheath and dissecting the posterior sheath between the internal oblique and transversus abdominis muscle.
  Interventions: Procedure: Posterior component separation technique.
- PCS without TAR (Active Comparator): by performing posterior component separation technique through inscion in the posterior rectus sheath and mesh placement in this plane without performing more advancement towards tranversus abdominis muscle.
  Interventions: Procedure: Posterior component separation technique.

INTERVENTIONS:
Procedure: Posterior component separation technique. — By dividing the posterior rectus sheath, a posterior plane is reached which can be advanced by dividing the transversus abdominis muscle with reinforcement of the midline with synthetic mesh.

SUMMARY:
* Assess short term outcome of posterior component separation technique(PCS) including the regain of the physiological function of the abdominal wall.
* Detect most common post operative complications related to AWR techniques in a 6 months duration after operation.

DETAILED DESCRIPTION:
posterior component separation(PCS) is one of the surgical techniques used in abdominal wall reconstruction plan foe management of relatively complex ventral hernia ,which cannot be treated with the conventional surgical way.

With or without transverses abdominis release(TAR) technique, (PCS) became widely accepted as surgical technique specially for large sized hernia defect, previous multiple laparotomies or unhealth abdominal soft tissue.

This study has a primary outcome which is detection of recurrence rate in patients under went posterior component separation technique in a period of 6 month after operation.

ELIGIBILITY:
Inclusion Criteria:

* patients with complex ventral hernia with contraindication to the conventional surgical therapy.

Exclusion Criteria:

1. patients with contraindication to long standing anesthesia.
2. patients with emergency hernia situation.
3. pregnant patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence | six month after operation
  develop ventral hernia recurrence

SECONDARY OUTCOMES:
post operative short term complications | One month after operation
  wound infection(hematoma, seroma) and wound dehiscence

CONTACTS AND LOCATIONS:
Overall Officials: Samir A Ammar, Study Director — Assiut University

REFERENCES:
- [Background] Ramirez OM, Ruas E, Dellon AL. "Components separation" method for closure of abdominal-wall defects: an anatomic and clinical study. Plast Reconstr Surg. 1990 Sep;86(3):519-26. doi: 10.1097/00006534-199009000-00023. PMID 2143588
- [Background] Novitsky YW, Elliott HL, Orenstein SB, Rosen MJ. Transversus abdominis muscle release: a novel approach to posterior component separation during complex abdominal wall reconstruction. Am J Surg. 2012 Nov;204(5):709-16. doi: 10.1016/j.amjsurg.2012.02.008. Epub 2012 May 16. PMID 22607741
- [Background] Kockerling F, Reinpold W, Schug-Pass C. [Abdominal wall hernias part 2 : Operative treatment techniques]. Chirurg. 2021 Aug;92(8):755-768. doi: 10.1007/s00104-021-01383-z. Epub 2021 Apr 1. German. PMID 33792765